CLINICAL TRIAL: NCT05038384
Title: Palliative, Rehabilitation, and Integrated Medicine Handbook for Self Care at Work Survey
Brief Title: Palliative, Rehabilitation, and Integrated Medicine Handbook for Self Care at Work
Status: Withdrawn | Type: Observational
Why Stopped: Accrual Limit
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0792; NCI-2021-08920 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0792 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-24; First posted 2021-09-09 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): Participants complete a survey over 20 minutes.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study investigates the usefulness of the Self Care at Work Handbook in order to generate an improved version. Information from this study may help researchers identify potential factors associated with perception and usefulness of the Self Care at Work Handbook.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the global perception of the perceived usefulness of the handbook, and the frequency that the handbook is consulted.

II. To explore the perceived usefulness of and adherence to each individual item of the handbook.

III. To solicit personnel for their ideas about the handbook, and particularly any additional handbook items they might suggest.

IV. To explore any relationships between the actual use or the perceived importance of each handbook item with respondents' self-reported professional satisfaction.

V. To explore any associations between responses to handbook items and professional, demographic, and work satisfaction characteristics before and during the coronavirus disease 2019 (COVID-19) crisis.

VI. To explore respondents' global perceptions of the usefulness and adherence to the handbook before and during the COVID-19 crisis.

OUTLINE:

Participants complete a survey over 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians in the Department of Palliative, Rehabilitation, and Integrative Medicine. This includes physicians, advanced practice providers (APPs), and other clinical staff in the Supportive Care Center and Acute Palliative Care Unit

Exclusion Criteria:

No

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinicians in the Department of Palliative, Rehabilitation, and Integrative Medicine at M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Global perception of usefulness | through study completion, an average of 1 year
  Will be assessed by survey question E, which has five options: very useful, useful, neither useful nor useless, useless and very useless. The main interest is the proportion of responders who select very useful and useful.
Frequency of consultation | through study completion, an average of 1 year
  Will be assessed by survey question D, which has five options: never, once a month or less, a few times a month, a few times a week and daily. The main interest is the proportion of responders who select daily and a few times a week.
Perceived usefulness of individual items | through study completion, an average of 1 year
  Will be assessed by survey question F 1-9. Frequency and proportion will be used to summarize each item. For responders who select neither useful nor useless, useless and very useless, additional questions about whether one item should be retained, discarded or modified will be summarized using frequency and proportion. Comments or suggestions will be collected for qualitative analysis.
Adherence to individual items | through study completion, an average of 1 year
  Will be assessed by survey question G 1-9. Frequency and proportion will be used to summarize each item. For responders who select neither useful nor useless, useless and very useless, additional questions about whether one item should be retained, discarded or modified will be summarized using frequency and proportion. Comments or suggestions will be collected for qualitative analysis.
Personal ideas about the handbook | through study completion, an average of 1 year
  Will be collected by survey question I and question J. Comments and suggestions will be collected and used to aggregate opinions toward handbook improvement.
Responders' self-reported professional satisfaction | through study completion, an average of 1 year
  Will be assessed by survey question K, L1, and L3. Association between the perceived usefulness and professional satisfaction will be evaluated by Chi-squared test or Fisher's exact test whichever appropriate. Association between the adherence and professional satisfaction will be evaluated by Chi-squared test or Fisher's exact test whichever appropriate.
Responders' profession | through study completion, an average of 1 year
  Will be summarized by survey question A, and responders' demographics will be summarized by survey question B and C. Responders' work satisfaction after coronavirus disease 2019 (COVID-19) will be examined by survey question L2 and L4. Association between the perceived usefulness and responders' profession/demographics/work satisfaction after COVID-19 will be evaluated by Chi-squared test or Fisher's exact test whichever appropriate. Association between the adherence and responders' profession/demographics/work satisfaction after COVID-19 will be evaluated by Chi-squared test or Fisher's exact test whichever appropriate.
Responders' global perceptions of usefulness and adherence to the handbook during COVID-19 | through study completion, an average of 1 year
  Will be assessed by survey question M, N and O, and frequency and proportion will be used to summarize the results.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bramati, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org